CLINICAL TRIAL: NCT02440152
Title: The Effectiveness of Deep Brain Stimulation for Opioid Relapse Prevention
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Suzhou Sceneray Medical Co. , Ltd (Industry); Shanghai Mental Health Center (Other); Institution of Neuroscience (Unknown); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Bomin Sun, Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-15
Record Dates: First submitted 2015-03-29; First posted 2015-05-12 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Opiate Addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep brain stimulation (Experimental)
  Interventions: Device: Suzhou Sceneray® DBS System

INTERVENTIONS:
Device: Suzhou Sceneray® DBS System — We plan to use the SceneRay 1242 (SceneRay, SuZhou, China) electrode with a diameter of 1.27 mm and 4 contacts. The SceneRay 1242 electrode combined with the SceneRay 1181 implantable pulse generator has the advantage of adaptive coverage area for the Ventral Capsule/Ventral Striatum, enabling simultaneous implantation in the nucleus accumbens (NAc; 2 ventral contacts) and the anterior limb of the internal capsule (ALIC; 2 dorsal contacts) with independently programmed parameters such as frequency, amplitude, and voltage; and remote and wireless programing, which allows for convenient and prompt adjustments in emergency situations. The contact length is 3.0 mm and the spacings between the ventral and dorsal contacts are 2 mm, 4 mm, and 4 mm, respectively, spanning a total length of 22.5 mm (3 + 2 + 3 + 4 + 3 + 4 + 3 mm, with 0.5 mm projecting from the electrode tip).

SUMMARY:
The nucleus accumbens (NAcc) has a significant role in the process of opiate addiction and the initiation of relapse after detoxification. There is evidence that deep brain stimulation (DBS) of the NAcc exerts a positive effect on individuals with severe heroin addiction via inhibitory action .

The investigators hypothesise that bilateral stimulation of the NAcc will significantly reduce withdrawal symptoms and thus enable the patients to substantially decrease their Levomethadone usage.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in Mandarin language
* Long lasting heroin addiction (determined by diagnostic-criteria in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition)
* Duration longer than 6 months
* A lack of response to long-term treatment
* Capacity to provide informed consent (understanding of the study purpose and methods)
* Substitution methadone treatment at a constant dose within three months prior to inclusion.

Exclusion Criteria:

* Clinical relevant psychiatric comorbidity (schizophrenic psychoses, bipolar affective diseases with psychotic symptoms)(MINI 6.0)
* Past stereotactic neurosurgical intervention
* Neurological disease (Abnormal PET-CT, MRI, EEG)
* Contraindications of MRI-examination, e.g. implanted cardiac pacemaker/ heart defibrillator
* Contraindications of stereotactic intervention, e.g. increased bleeding-disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases)
* Serious and unstable organic diseases (e.g. unstable coronal heart disease)
* HIV positive
* Pregnancy and/or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Weekly urine tests | Baseline (preoperative), 3 months, 6 months, 9 months, 12 months, 18 months, 24 months

SECONDARY OUTCOMES:
Change in 10-point visual analog scale (VAS) craving score for opioid drugs | Baseline (preoperative), 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
Change in Hamilton Anxiety Scale | Baseline (preoperative), 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
Change in Hamilton Depression Scale-17 | Baseline (preoperative), 3 months, 6 months, 9 months, 12 months, 18 months, 24 months
Change in SF-36 assessment | Baseline (preoperative), 6 months, 12 month, 24 month
Neuropsychological measures（Scores of Iowa gambling task and Model task） | Baseline (preoperative), Intraoperative,6 months,12month,24month

CONTACTS AND LOCATIONS:
Overall Officials: Bomin Sun, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Shanghai RuiJin Hospital Psychitric Department, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luigjes J, van den Brink W, Feenstra M, van den Munckhof P, Schuurman PR, Schippers R, Mazaheri A, De Vries TJ, Denys D. Deep brain stimulation in addiction: a review of potential brain targets. Mol Psychiatry. 2012 Jun;17(6):572-83. doi: 10.1038/mp.2011.114. Epub 2011 Sep 20. PMID 21931318
- [Result] Kuhn J, Moller M, Treppmann JF, Bartsch C, Lenartz D, Gruendler TO, Maarouf M, Brosig A, Barnikol UB, Klosterkotter J, Sturm V. Deep brain stimulation of the nucleus accumbens and its usefulness in severe opioid addiction. Mol Psychiatry. 2014 Feb;19(2):145-6. doi: 10.1038/mp.2012.196. Epub 2013 Jan 22. No abstract available. PMID 23337942
- [Result] Valencia-Alfonso CE, Luigjes J, Smolders R, Cohen MX, Levar N, Mazaheri A, van den Munckhof P, Schuurman PR, van den Brink W, Denys D. Effective deep brain stimulation in heroin addiction: a case report with complementary intracranial electroencephalogram. Biol Psychiatry. 2012 Apr 15;71(8):e35-7. doi: 10.1016/j.biopsych.2011.12.013. Epub 2012 Jan 26. No abstract available. PMID 22281120
- [Result] Zhou H, Xu J, Jiang J. Deep brain stimulation of nucleus accumbens on heroin-seeking behaviors: a case report. Biol Psychiatry. 2011 Jun 1;69(11):e41-2. doi: 10.1016/j.biopsych.2011.02.012. Epub 2011 Apr 13. No abstract available. PMID 21489407